### **Statistical Analysis Plan (SAP)**

**Title:** Statistical Analysis Plan for "The Effect of Experiential Learning-Based First-aid Training on Knowledge and Self-efficacy of Parents of Children with Intellectual Disabilities" **Objectives:** To assess changes in first-aid knowledge, To assess changes in first-aid self-efficacy.

### **Analysis Populations:**

Full Analysis Set (FAS): All randomized participants who completed pre- and post-tests.

Per Protocol (PP): Participants who attended all four training sessions (intervention group).

#### **Statistical Methods:**

**Descriptive Statistics:** Mean, standard deviation, frequency, and percentages for sociodemographic and baseline variables.

**Baseline Comparisons:** Chi-square test (categorical variables), independent samples t-test (continuous variables).

# **Primary Outcome Analysis:**

Knowledge scores: Comparison of pre- and post-test scores within groups (paired t-test). Between-group differences in change scores: Independent t-test.

# **Secondary Outcome Analysis:**

Self-efficacy scores: Same method as knowledge scores.

**Effect Size:** Cohen's d will be calculated to estimate the magnitude of the intervention effect.

**Assumptions Check:** Normality (skewness, kurtosis). Non-normal data will be analyzed with non-parametric equivalents (Wilcoxon signed-rank, Mann–Whitney U).

**Significance Level:** p < 0.05, two-tailed.

**Software:** SPSS Statistics v25, G\*Power 3.1.9.7 for sample size